CLINICAL TRIAL: NCT06736457
Title: Study on Safety and Performance of AdvanCore Bone Void Filler
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Artur Salgado SA (Industry)
Collaborators: NAMSA (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ADV-01
Record Dates: First submitted 2024-12-11; First posted 2024-12-16 (Actual); Last update posted 2025-05-31 (Actual); Status verified 2025-05

CONDITIONS: Bone Fractures; Bone Defects; Bone Loss; Bone Graft
Keywords: Bone graft; Bone substitute; Bone regeneration; AdvanCore; Beta-Tricalcium Phosphate; Synthetic bone graft
MeSH Terms: conditions — Fractures, Bone; Bone Diseases, Metabolic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Long-bone injuries (Experimental): Group formed by subjects with long-bone injuries treated using AdvanCore blocks, wedges, or granules.
  Interventions: Procedure: AdvanCore bone grafting
- Spine injuries (Experimental): Group formed by subjects with spine injuries treated using AdvanCore granules.
  Interventions: Procedure: AdvanCore bone grafting
- Maxillofacial injuries (Experimental): Group formed by subjects with maxillofacial injuries treated using AdvanCore granules.
  Interventions: Procedure: AdvanCore bone grafting

INTERVENTIONS:
Procedure: AdvanCore bone grafting — AdvanCore medical device is implanted making sure that is in direct contact with all surfaces of the defect area.

SUMMARY:
The objective of this study is to evaluate the safety and performance of AdvanCore implantable bone graft through a 12-month follow-up period in a prospective, parallel-group design, non-controlled, open label, multi-center and real-world setting study. This study is intended to satisfy post-market clinical follow-up requirements of CE Mark in Europe.

DETAILED DESCRIPTION:
AdvanCore is a porous beta-tricalcium phosphate CE-marked medical device. It is intended to be used to aid in the bone regeneration process in situations where bone is damaged beyond the limits of its self-healing ability. The target population is constituted by adult subjects in need of bone grafting of mechanically unaffected, pathologic, or traumatic bone defects caused by surgery or trauma.

AdvanCore is produced in the shape of blocks, wedges, or granules in different sizes and is surgically placed into spaces between or around broken bone (fractures) or in holes (defects). The site to be augmented must be free from infection and free from soft or granulation tissue. AdvanCore must contact cancelous bone and may be pressed into the defect area by hand or shaped more accurately to fit the area. It can be used as is, impregnated with subjects' blood/ bone marrow and/ or mixed with medicinal substances under the responsibility of the qualified professionals.

AdvanCore acts as a temporary scaffold and is not intended to provide mechanical support during the healing process. Additional therapy for load-bearing (such as osteosynthesis) is indicated if the bone does not comply with the required biomechanical function.

The study on safety and performance of AdvanCore bone void filler will be conducted in European sites and include up to 190 subjects requiring bone implant surgery, which will be divided in 3 different groups:

* Group 1- This group is formed by those subjects with long-bone injuries. The treatment of this type of lesion may be performed using blocks, wedges, or granules.
* Group 2- Subjects included in this group suffer from spine injuries, which can be treated using granules.
* Group 3- Those subjects with maxillofacial injuries are included in this group. In this case, granules are used to treat the lesion.

The primary safety endpoint of this study is defined as freedom of bone reintervention due to AdvanCore usage at 6 months, analyzing the occurrence of Adverse Events or Serious Adverse Events [(S)AEs] related to the device usage and/ or AdvanCore procedure that may lead to subjects' reoperation.

The primary performance endpoint will analyze the AdvanCore osteointegration after 6 months of surgery, studying the percentage of subjects with successful osteointegration at the defined time point. AdvanCore will be considered successfully osteointegrated when no presence of fibrotic tissue surrounding the implant is detected.

Secondary endpoints planned for this clinical investigation are listed below:

* Evaluation of (S)AEs related to the procedure;
* Evaluation of (S)AEs related to the device;
* Freedom of reintervention due to AdvanCore usage;
* AdvanCore osteointegration;
* AdvanCore resorption rate, assessed as the percentage of subjects with successful bone graft resorption.

The clinical investigation has been designed to involve as little pain, discomfort, fear, and any other foreseeable risk as possible for subjects.

ELIGIBILITY:
Inclusion Criteria:

* Adult subjects ≥ 18 years old, male or female.
* Subjects who are eligible for a bone grafting/bone void filler procedure.
* Subjects with bone lesions beyond the limits of the bone's self-healing ability.
* Subjects, and/or an authorized representative, who are willing and capable of providing informed consent, participating in all testing associated with this clinical investigation at an approved clinical investigational center.
* Subjects with only one fracture susceptible to treatment with an AdvanCore implant.

Exclusion Criteria:

* Subjects with any AdvanCore contraindication for implantation or use.
* Subjects with hypersensitivity to any of the AdvanCore components.
* Subjects with infections or soft/granulation tissue in the area to place bone graft.
* Subjects who are currently enrolled in another investigational study or registry that would directly interfere with the current study.
* Women who are breastfeeding or of childbearing potential who are, or plan to become, pregnant during the time of the study (method of assessment upon physician's discretion).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 190 (Estimated)
Dates: Start 2025-05-29 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Freedom of bone reintervention (safety) | 6 months post-surgery
  The primary safety endpoint is defined as freedom of bone reintervention due to AdvanCore usage at 6 months, analyzing the occurrence of (S)AEs related to the device usage and/ or AdvanCore procedure that may lead to subjects' reoperation.
Successful osteointegration (performance) | 6 months post-surgery
  The primary performance endpoint will analyze the AdvanCore integration at 6 months of surgery. This process is defined as osteointegration, which refers to the direct structural and functional connection of the living bone with the surface of the implant. The implant osteointegration will be assessed by imaging techniques selected according to the current clinical practices of each site. In this regard, the primary performance endpoint will be analyzed by considering the percentage of subjects with successful osteointegration at the defined timeline. AdvanCore will be considered successfully osteointegrated when the presence of fibrotic tissue surrounding the implant is not detected.

SECONDARY OUTCOMES:
Evaluation of Adverse Events or Serious Adverse Events [(S)AEs] related to the procedure (safety) | 30-days post-surgery
  Record of Adverse Events or Serious Adverse Events [(S)AEs] related to the procedure during a 12-month follow-up period. In all cases, the analysis population will be the Per-Protocol population, and results will be presented as the incidence (in percentage) of (S)AEs, with a 95% confidence.
Evaluation of (S)AEs related to the procedure (safety) | 3 months post-surgery
  Record of (S)AEs related to the procedure during a 12-month follow-up period. In all cases, the analysis population will be the Per-Protocol population, and results will be presented as the incidence (in percentage) of (S)AEs, with a 95% confidence.
Evaluation of (S)AEs related to the procedure (safety) | 6 months post-surgery
  Record of (S)AEs related to the procedure during a 12-month follow-up period. In all cases, the analysis population will be the Per-Protocol population, and results will be presented as the incidence (in percentage) of (S)AEs, with a 95% confidence.
Evaluation of (S)AEs related to the procedure (safety) | 12 months post-surgery
  Record of (S)AEs related to the procedure during a 12-month follow-up period. In all cases, the analysis population will be the Per-Protocol population, and results will be presented as the incidence (in percentage) of (S)AEs, with a 95% confidence.
Evaluation of (S)AEs related to the device (safety) | 30 days post-surgery
  Record of (S)AEs related to the device during a 12-month follow-up period. In all cases, the analysis population will be the Per-Protocol population, and results will be presented as the incidence (in percentage) of (S)AEs, with a 95% confidence.
Evaluation of (S)AEs related to the device (safety) | 3 months post-surgery
  Record of (S)AEs related to the device during a 12-month follow-up period. In all cases, the analysis population will be the Per-Protocol population, and results will be presented as the incidence (in percentage) of (S)AEs, with a 95% confidence.
Evaluation of (S)AEs related to the device (safety) | 6 months post-surgery
  Record of (S)AEs related to the device during a 12-month follow-up period. In all cases, the analysis population will be the Per-Protocol population, and results will be presented as the incidence (in percentage) of (S)AEs, with a 95% confidence.
Evaluation of (S)AEs related to the device (safety) | 12 months post-surgery
  Record of (S)AEs related to the device during a 12-month follow-up period. In all cases, the analysis population will be the Per-Protocol population, and results will be presented as the incidence (in percentage) of (S)AEs, with a 95% confidence.
Freedom of reintervention (safety) | 12 months post-surgery
  Freedom of reintervention due to AdvanCore usage, analyzing the occurrence of (S)AEs related to the device usage and/ or AdvanCore procedure that may lead to subjects' reoperation.
Successful osteointegration (performance) | 30 days post-surgery
  The implant osteointegration will be assessed by imaging techniques selected according to the current clinical practices of each site. This analysis will determine the percentage of number of subjects with successful implant osteointegration. AdvanCore will be considered successfully osteointegrated when the presence of fibrotic tissue surrounding the implant is not detected.
Successful osteointegration (performance) | 3 months post-surgery
  The implant osteointegration will be assessed by imaging techniques selected according to the current clinical practices of each site. This analysis will determine the percentage of number of subjects with successful implant osteointegration. AdvanCore will be considered successfully osteointegrated when the presence of fibrotic tissue surrounding the implant is not detected.
Successful osteointegration (performance) | 12 months post-surgery
  The implant osteointegration will be assessed by imaging techniques selected according to the current clinical practices of each site. This analysis will determine the percentage of number of subjects with successful implant osteointegration. AdvanCore will be considered successfully osteointegrated when the presence of fibrotic tissue surrounding the implant is not detected.
Successful resorption (performance) | 6 months post-surgery
  Resorption is the breakdown and assimilation of the implant in the cycle of bone growth. The implant resorption will be assessed by imaging techniques selected according to the current clinical practices of each site. This analysis will determine the percentage of number of subjects with successful implant resorption. The successful resorption rate will be reached if at least 25% of the AdvanCore graft cannot be detected at 6 months.
Successful resorption (performance) | 12 months post-surgery
  Resorption is the breakdown and assimilation of the implant in the cycle of bone growth. The implant resorption will be assessed by imaging techniques selected according to the current clinical practices of each site. This analysis will determine the percentage of number of subjects with successful implant resorption. The successful resorption rate will be reached if at least 50% of the AdvanCore graft cannot be detected at 12 months.

CONTACTS AND LOCATIONS:
Locations (4):
- Portugal (4):
  - Unidade Local de Saúde do Alto Ave, Guimarães, Braga District
  - Unidade Local de Saúde de São João, Porto, Porto District
  - Unidade Local de Saúde do Médio Tejo, Tomar, Santarém District
  - Unidade Local de Saúde de Trás-os-Montes e Alto Douro, Lordelo, Vila Real District

IPD SHARING:
Plan to Share IPD: No